CLINICAL TRIAL: NCT03152253
Title: Live Inspired: Individually Tailored and Integrated Social Support Network for Tobacco Cessation
Brief Title: Individually Tailored and Integrated Social Support Network for Tobacco Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: Live Inspired, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 860485-7
Record Dates: First submitted 2017-05-11; First posted 2017-05-12 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-03

CONDITIONS: Smoking Cessation
Keywords: Tobacco, Smoking, Text Message
MeSH Terms: conditions — Smoking Cessation; Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Text Message for Smoking Cessation (Experimental): smoking cessation promotion messages and medication reminders sent via text messages for up to 30 days before quit day and 8 weeks following quit day, along with access to a social support chat room
  Interventions: Behavioral: Text My Quit (TMQ); Behavioral: Peer Support
- Non-Interventional Text Messages (Placebo Comparator): General motivational text messages sent on the same schedule at TMQ arm of the study with access to a social support chat room.
  Interventions: Behavioral: Peer Support; Other: Motivational Messages

INTERVENTIONS:
Behavioral: Text My Quit (TMQ) — Text messages designed to aid smoking cessation
  Arms: Text Message for Smoking Cessation
Behavioral: Peer Support — A group chat room for peer support
Other: Motivational Messages — Generic motivational messages not related to smoking cessation
  Arms: Non-Interventional Text Messages

SUMMARY:
This study will continue development of a quit smoking program delivered through text messaging. Upon completion of programming we will enroll 280 participants and randomize them to a control condition or the intervention condition. Assessments will occur at enrollment, and both 3 and 6 month follow ups.

DETAILED DESCRIPTION:
This study builds on pilot work in which Live Inspired LLC and research partners developed T2Q (formerly "Text-2-Quit") a smoking cessation intervention delivered through text messaging. T2Q is a unique program with a number of features that provide superior support and service compared to existing text message quit smoking products. T2Q is 100% accessible through text messaging provides medication support for quitting smoking, an integrated social support network and live counseling. This phase II project will add functionality to accommodate use of multiple forms of quit smoking medications, and then conduct a rigorous test of the efficacy of T2Q among 280 adult smokers and examine smoking outcomes compared to controls at 3 and 6 months follow up. The study will also examine changes in smoking-related attitudes and behaviors among T2Q users to identify strengths and any potential weaknesses that may affect T2Q's impact on smoking outcomes. Analyses will examine the quality of social interactions within the T2Q integrated social support network and their role in promoting smoking abstinence. We will also conduct interviews with study participants in the T2Q arm to enable understanding of the user's experience with T2Q. Results of this trial will demonstrate the efficacy of T2Q - providing important credibility needed for successful commercialization. This research will also provide important data for possible enhancements to improve consumer appeal prior to commercialization.

This proposal finalizes development and testing of a unique, highly scalable intervention that can reach a U.S. market comprised of over 34 million adult smokers who use text messaging, and provide them with effective, evidence-based treatment. Text messaging enjoys near-market saturation and is a widely preferred method of communication with deep penetration across diverse groups. Wide availability of an attractive and effective smoking cessation program such as T2Q, may exert a powerful, sustained impact on public health

ELIGIBILITY:
Inclusion Criteria:

* age >18
* current daily cigarette smoker
* use of text messaging at least once per week
* interested in quitting smoking within the next 30 days
* has access to a physician or healthcare provider
* no current drug/alcohol abuse.

Exclusion Criteria:

* Non-English Speaking
* Currently using quit-smoking medications or therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Smoking Abstinence | 6 month follow up
  Self-report of no smoking for the past 7 days

SECONDARY OUTCOMES:
Social support network use | 12 weeks
  number of messages sent to the chat room

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Deutsch, BS, Principal Investigator — Live Inspired, LLC
Locations (1):
- The Miriam Hospital- CORO building, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bock BC, Rosen RK, Barnett NP, Thind H, Walaska K, Foster R, Deutsch C, Traficante R. Translating Behavioral Interventions Onto mHealth Platforms: Developing Text Message Interventions for Smoking and Alcohol. JMIR Mhealth Uhealth. 2015 Feb 24;3(1):e22. doi: 10.2196/mhealth.3779. PMID 25714907